CLINICAL TRIAL: NCT06194331
Title: Optimizing Suicide Prevention Strategies for Pediatric Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Pediatric Research in Office Settings (Network); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephanie Stepp, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY23040042; 1R34MH132932-01 (NIH)
Record Dates: First submitted 2023-11-30; First posted 2024-01-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Suicidal Ideation; Suicidal and Self-injurious Behavior; Depression
Keywords: Suicidal Ideation; Suicidal and Self-injurious Behavior; Depression
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study will utilize a stepped wedge design in which 4 PROS practices start with usual care initially and are randomly chosen to transition to iCHART-cASAP at different times in such a way as half of the participants will receive TAU and half will receive iCHART-cASAP. All sites will be initially monitored for at least 3 months during TAU. This will be followed by a staggered adoption of iCHART-cASAP. At each time period, a new site will begin implementing the intervention. Block randomization determines the order each site begins the intervention phase. Each time period (approximately 3 months), a web-based system will be used to assign the next clinic to begin using iCHART-cASAP. Research staff will be available to assist with consenting participants and assisting with study procedures.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor and the investigator will be blinded to whether or not the participant received the iCHART/cASAP intervention or if they are receiving treatment as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCHART/cASAP (Experimental): An intervention previously studied in the ETUDES Center along with a computerized version of our As Safe As Possible intervention.
  1. Safety Planning App for suicidal youth which enables a primary care provider to streamline the gold standard of care for those with current suicidality symptoms through an app;
  2. Mental Health Screener questionnaire that gathers additional mental health symptoms, treatment preferences, and family's readiness for treatment engagement to help a primary care provider make a personalized, tailored treatment plan a suicidal youth is more likely to adhere to;
  3. Text Messages which aims to provide texts for 2-3 weeks to motivate you to engage with the safety plan and recommended treatment following the patient visit.
  4. cASAP is a computerized version of the As Safe As Possible intervention that offers self-led modules with psychoeducation about safety planning, cognitive-behavioral skills to cope with distress, and facilitate collaboration with parents.
  Interventions: Behavioral: iCHART/cASAP
- Treatment as usual (Active Comparator): When patients disclose suicidal ideation on the PHQ-9, a treatment as usual approach will be given to the patient and their parent by the pediatrician which includes a paper safety plan will be completed and given to the patient and a referral placed for the patient to begin behavioral health services.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: iCHART/cASAP — When patients disclose suicidal ideation on the PHQ-9, the intervention of iCHART/cASAP will be implemented in the pediatrician's office, and in collaboration with parents, which includes safety planning, teaching skills to improve distress tolerance and emotion regulation all on the teen's smart device. iCHART/cASAP will include: Screening Wizard, a digital screening tool that will guide the provider to gauge patient satisfaction with current treatment and making further personalized treatment recommendations; cASAP, a computerized version of the As Safe As Possible intervention that focuses on psychoeducation in safety planning, distress tolerance, and emotion regulation skills; BRITE, a safety planning app with distress monitoring that a teen can be guided through with automated onboarding manuals; Text2Connect, an automated text messaging sent centrally to patients and parents to enhance treatment adherence.
  Arms: iCHART/cASAP
Behavioral: Treatment as usual — When patients disclose suicidal ideation on the PHQ-9, a treatment as usual approach will be given to the patient and their parent by the pediatrician which includes a paper safety plan will be completed and given to the patient and a referral placed for the patient to begin behavioral health services.
  Arms: Treatment as usual

SUMMARY:
Increasing rates of suicidal thoughts and behaviors among adolescents must be addressed. The study will adapt and collect preliminary effectiveness data on a digital suicide prevention intervention that can be delivered in pediatric primary care settings by front line pediatricians. The study has the potential to offer a low-cost and scalable primary care intervention that may decrease risk of suicide among at-risk youth.

DETAILED DESCRIPTION:
The study proposed is a treatment development study to enhance the capacity of pediatric primary care (PPC) to identify and manage suicidal youth by adapting iCHART for PPC settings that lack onsite behavioral health (BH) providers.

Stepped Wedge Cluster Randomized Pilot Trial: Conduct a stepped wedge cluster randomized pilot trial of iCHART-cASAP vs. usual care across 4 PROS practices (across urban, suburban, and rural settings). Up to 20 providers (up to 5 providers per practice) will be enrolled. Following a 3-month baseline period when all practices provide usual care, practices will be randomized to onset to offering the intervention at one of the four, 3-month intervention onset intervals. Each practice will enroll a total of 15 youth across the 15-month pilot trial period for a total of 60 youth. 30 youth will receive usual care and 30 youth will receive iCHART-cASAP.

Delivery of Intervention Intervention will be delivered to adolescent patients and their caregivers receiving services at pediatric primary care practices within the PROS network.When PPC providers are assigned to the usual condition, patients will receive usual practices following identification of suicide risk on the PHQ-9-M. When PPC providers have crossed over to the iCHART- cASAP intervention condition, patients who are identified as suicidal will receive links from PPC providers/office staff to complete cASAP + onboard BRITE app to receive the safety planning and skills training intervention for adolescent and parent/caregiver. Once that is completed, PPC providers receive a summary report and review the safety plan with the patient and parent/caregiver, making revisions as needed. The provider then reviews treatment plan, including behavioral health referrals and schedules follow-up appointment. Next, the PPC provider/office staff enters referral recommendations and follow-up appointment reminders into iCHART's Text2Connect feature, which will increase engagement with the safety plan and facilitate adherence with treatment recommendations.

Providers will approach patients and parents/caregivers about the research study during their office visit, and interested families will complete a permission to contact form for research staff. Research staff will contact and describe the study, answer any questions, and obtain parental consent/youth assent.

Sample Size and Power Considerations Once usability testing is complete, 60 participants will be recruited from 4 practices randomized to begin utilizing iCHART during one of the 3-month intervention intervals. At the end of the trial, 30 participants will be enrolled when practices were delivering usual care and 30 participants will be enrolled when practices were delivering iCHART- cASAP.

Sample size and power considerations center on the precision of confidence interval (CI) width estimation for feasibility outcomes. Based on best practices for feasibility studies, and given the sample size of 60 and 5% type I error rate, there is ability to estimate 95% confidence interval with margin-of-errors ≤0.33 for the primary outcomes of depression and suicidal thoughts and behaviors.

ELIGIBILITY:
Youth Inclusion:

* 12-17 years old
* Parent/legal guardian consents for youth to be in study
* English fluency and literacy-own a smart phone or device
* PHQ-9M score indicating moderate or severe depression or suicidal ideation in past month, past 2 weeks, or an attempt in their lifetime

Caregiver/Parent inclusion:

-English fluency and literacy

Youth Exclusion:

* evidence of intellectual delay
* pervasive developmental disorder
* other condition from medical history that would prohibit comprehension of questions or modules

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation and behavior on PHQ-9M | Baseline
  Suicidal ideation and attempt will be measured by 3 items on the PHQ-9-M (item #9 with scaled options of '0=not at all, 1=several days, 2=more than half the days, 3=nearly every day', past month ideation, prior suicide attempt) as a primary outcome.
Suicidal ideation and behavior on PHQ-9M | 1-month follow-up
  Suicidal ideation and attempt will be measured by 3 items on the PHQ-9-M (item #9 with scaled options of '0=not at all, 1=several days, 2=more than half the days, 3=nearly every day', past month ideation, prior suicide attempt) as a primary outcome.
Suicidal ideation and behavior on PHQ-9M | 3-month follow-up
  Suicidal ideation and attempt will be measured by 3 items on the PHQ-9-M (item #9 with scaled options of '0=not at all, 1=several days, 2=more than half the days, 3=nearly every day', past month ideation, prior suicide attempt) as a primary outcome.
Suicidal ideation and behavior on PHQ-9M | 6-month follow-up
  Suicidal ideation and attempt will be measured by 3 items on the PHQ-9-M (item #9 with scaled options of '0=not at all, 1=several days, 2=more than half the days, 3=nearly every day', past month ideation, prior suicide attempt) as a primary outcome.
Suicidal ideation and behavior on CSSRS | Baseline
  Suicidal attempt & ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). Assign score of 0 if no ideation/behavior present and assign a score of 1 if ideation/behavior present. A "yes" answer any time during treatment to question 9 on the PHQ-9 indicates suicidal ideation. A "yes" answer any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 7-10) on the C-SSRS. C-SSRS Categories 7-10 are as follows: 7-Aborted Attempt 8-Interrupted Attempt 9-Actual Attempt (non-fatal) 10-Completed Suicide. Any score greater than 0 is important/may indicate need for intervention.
Suicidal ideation and behavior on CSSRS | 1-month follow-up
  Suicidal attempt & ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). Assign score of 0 if no ideation/behavior present and assign a score of 1 if ideation/behavior present. A "yes" answer any time during treatment to question 9 on the PHQ-9 indicates suicidal ideation. A "yes" answer any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 7-10) on the C-SSRS. C-SSRS Categories 7-10 are as follows: 7-Aborted Attempt 8-Interrupted Attempt 9-Actual Attempt (non-fatal) 10-Completed Suicide. Any score greater than 0 is important/may indicate need for intervention.
Suicidal ideation and behavior on CSSRS | 3-month follow-up
  Suicidal attempt & ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). Assign score of 0 if no ideation/behavior present and assign a score of 1 if ideation/behavior present. A "yes" answer any time during treatment to question 9 on the PHQ-9 indicates suicidal ideation. A "yes" answer any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 7-10) on the C-SSRS. C-SSRS Categories 7-10 are as follows: 7-Aborted Attempt 8-Interrupted Attempt 9-Actual Attempt (non-fatal) 10-Completed Suicide. Any score greater than 0 is important/may indicate need for intervention.
Suicidal ideation and behavior on CSSRS | 6-month follow-up
  Suicidal attempt & ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). Assign score of 0 if no ideation/behavior present and assign a score of 1 if ideation/behavior present. A "yes" answer any time during treatment to question 9 on the PHQ-9 indicates suicidal ideation. A "yes" answer any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 7-10) on the C-SSRS. C-SSRS Categories 7-10 are as follows: 7-Aborted Attempt 8-Interrupted Attempt 9-Actual Attempt (non-fatal) 10-Completed Suicide. Any score greater than 0 is important/may indicate need for intervention.
Depression Severity | Baseline
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity, as a primary outcome. The PHQ-9M uses scaled responses of '0=not at all, 1=several days, 2=more than half the days, 3=nearly every day'.
Depression Severity | 1-month follow-up
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity, as a primary outcome. The PHQ-9M uses scaled responses of '0=not at all, 1=several days, 2=more than half the days, 3=nearly every day'.
Depression Severity | 3-month follow-up
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity, as a primary outcome. The PHQ-9M uses scaled responses of '0=not at all, 1=several days, 2=more than half the days, 3=nearly every day'.
Depression Severity | 6-month follow-up
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity, as a primary outcome. The PHQ-9M uses scaled responses of '0=not at all, 1=several days, 2=more than half the days, 3=nearly every day'.
Application utilization | Monitored over 6 months
  Use of the iCHART-cASAP components and web portals will be monitored. Utilization will be measured by the number and proportion of adolescents, parents, and providers who have engaged with the application over time.
Service Utilization - SACA | Baseline
  Frequency and type of behavioral/mental health and primary care services using the Service Assessment for Children and Adolescents (SACA).
Service Utilization - SACA | 6-month follow-up
  Frequency and type of behavioral/mental health and primary care services using the Service Assessment for Children and Adolescents (SACA).
Patient Satisfaction | 6-month follow-up
  Satisfaction will be measured with the Client Satisfaction Questionnaire (CSQ). The scaled options for the CSQ vary as follows:
  Question 1: "4=Excellent, 3=Good, 2=Fair, 1=Poor" Question 2: "1=No, Definitely Not, 2=No, Not Really, 3=Yes, Generally, 4=Yes, Definitely" Question 3: "4=Almost all of my needs have been met, 3=Most of my needs have been met, 2=Only a few of my needs have been met, 1=None of my needs have been met" Question 4: "1=No, definitely not, 2=No, I don't think so, 3=Yes, I think so, 4=Yes, Definitely" Question 5: "1=Quite Dissatisfied, 2=Indifferent or mildly dissatisfied, 3=Mostly satisfied, 4=Very satisfied" Question 6: "4=Yes, they helped a great deal, 3=Yes, they helped somewhat, 2=No, they really didn't help, 1=No, they seemed to make things worse" Question 7: "4=Very satisfied, 3=Mostly satisfied, 2=Indifferent or mildly dissatisfied, 1=Quite dissatisfied" Question 8: "1=No, Definitely not, 2=No, I don't think so, 3=Yes, I think so, 4=Yes, Definitely
Acceptability | 6-month follow-up
  Acceptability of cASAP and the iCHART-cASAP intervention will be assessed through the Acceptability of Intervention Measure (AIM). The scaled options for the measure are: '1=Completely disagree, 2=Disagree, 3=Neither agree nor disagree, 4=Agree, 5=Completely agree'
Patient Usability | 6-month follow-up
  Patient usability will be measured by the Systems Usability Survey (SUS). The System Usability Scale uses scaled options of: '1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree'.
Provider Feasibility of Intervention Measure | 6-month follow-up
  Provider Feasibility will be measured using the Feasibility of Intervention Measure (FIM). The Feasibilty of Intervention Measure uses scaled options of: '1=Completely disagree, 2=Disagree, 3=Neither agree nor disagree, 4=Agree, 5=Completely agree'.
Provider Usability | 6-month follow-up
  System Usability Scale (SUS) will assess usability. The System Usability Scale uses scaled options of: '1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree'.

SECONDARY OUTCOMES:
Stress | Baseline
  Stress will be measured by the Pediatric Patient-Reported Outcomes Measurement Information System (PROMIS) Psychological Stress Experiences 4- item Short Form. The scaled options for this measure are: '1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always'.
Stress | 1-month follow-up
  Stress will be measured by the Pediatric Patient-Reported Outcomes Measurement Information System (PROMIS) Psychological Stress Experiences 4- item Short Form. The scaled options for this measure are: '1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always'.
Stress | 3-month follow-up
  Stress will be measured by the Pediatric Patient-Reported Outcomes Measurement Information System (PROMIS) Psychological Stress Experiences 4- item Short Form. The scaled options for this measure are: '1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always'.
Stress | 6-month follow-up
  Stress will be measured by the Pediatric Patient-Reported Outcomes Measurement Information System (PROMIS) Psychological Stress Experiences 4- item Short Form. The scaled options for this measure are: '1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always'.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Stepp, Principal Investigator — University of Pittsburgh
Locations (1):
- Pediatric Research in Office Settings National Headquarters, Itasca, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the NIMH's data sharing and data use policies this research study and clinical trial will be compliant with requirements for depositing data with the NIMH Data Archive (NDA) in the National Database for Clinical Trials Related to Mental Illness (NDCT). Specific statements will be added to the consent forms to allow for data sharing. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study staff will work to create unique identifiers for all participants, create a data dictionary for all variables, and submit raw data bi-annually. Data will be released to NDCT after manuscripts reporting primary findings are accepted for publication.
Access Criteria: In addition to public access to the NDCT, data can be accessed by contacting study investigators.
URL: http://nda.nih.gov

DOCUMENTS (2):
  • Study Protocol (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT06194331/Prot_000.pdf
  • Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT06194331/ICF_001.pdf